CLINICAL TRIAL: NCT01073215
Title: Primary Care Research Network for the Treatment of Adolescent Obesity
Acronym: TEENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Pennsylvania Department of Health (Other Government); Geisinger Clinic (Other); University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-005084; SAP4100033130
Record Dates: First submitted 2010-02-19; First posted 2010-02-23 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Obesity
Keywords: Adolescents; Obesity; Weight Management; Family-based Lifestyle Modification
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group Condition (Active Comparator)
  Interventions: Behavioral: Family-Based Lifestyle Modification Program
- Self-Guided Condition (Experimental)
  Interventions: Behavioral: Family-Based Lifestyle Modification

INTERVENTIONS:
Behavioral: Family-Based Lifestyle Modification — The Self-Guided condition will receive the same manual content and recommendations for eating and physical activity as the Group Condition. Since this approach is primarily home-based, participants in this condition will also receive additional tips and guidelines to assist the family in following the program at home. There will be 6 visits with the health coach at weeks 01, 04, 08, 24, 40, and 52. Participants will receive 2 phone calls from health coach at weeks 16 and 32. Parents and teens will be encouraged to hold weekly meetings at home to discuss program goals and progress.
  Other Names: TEENS Study
  Arms: Self-Guided Condition
Behavioral: Family-Based Lifestyle Modification Program — The Group condition will consist of a comprehensive family based lifestyle modification program of 23 visits (8 weekly, 8 bi-weekly, 7 monthly).
  Intervention visits include a combination of 17 group sessions and 6 individual meetings with health coach. There will be 7 phone calls two weeks after each monthly visit. Adolescents and their parents attend concurrent group meetings. The content of the sessions will include topics related to nutrition, physical activity, and behavior modification for weight management.
  Other Names: TEENS Study
  Arms: Group Condition

SUMMARY:
The "Primary Care Research Network for the Treatment of Adolescent Obesity" will establish infrastructure within the primary care setting to support programmatic research on weight loss for underserved adolescents, primarily urban African Americans, rural Caucasians, and Latinos. Using primary care settings, to which many youths already have entry, may increase access for underserved adolescents to participate in obesity treatment and research. The primary project will be a 12 month randomized controlled study comparing the relative effectiveness of two interventions for weight reduction: Group Condition (a family based lifestyle modification program delivered by health care providers in 23 sessions); Self-Guided Condition (a family based lifestyle modification program that combines a self-guided, home-based approach with 6 sessions delivered by health care providers).

DETAILED DESCRIPTION:
The broad objective is to establish a Center of Excellence for Research on Obesity at The Children's Hospital of Philadelphia (CHOP) that will create a statewide, collaborative research network to develop and test effective treatments for reducing adolescent obesity and related medical co-morbidities in underserved populations. Collaborating institutions include Lincoln University (LU), Geisinger Health System (GHS), and the University of Pennsylvania (UPenn). Given the locations of these institutions, we will focus on urban African Americans and Latinos and rural Caucasian adolescents. The novelty of this program will be the use of a family-based, lifestyle modification program within the pediatric primary care setting with interdisciplinary teams trained to treat obese adolescents. Specific aims are to: a) design, implement, and evaluate improved treatments for obese teenagers, b) conduct focus groups and treatment development projects to better understand the needs of these populations and c) train, minority students and faculty to become healthcare research professionals. The primary research project will be a randomized clinical trial occurring at two sites: CHOP and GHS. In a four-year study, 156 adolescents (ages 12-16) will be randomized to either a one-year, 23 session, multi-family, group based Lifestyle Modification Program known as the Group Condition, or to a one-year, six-session Self-Guided Condition. Both Group and Self-Guided will be tested as possible treatment protocols for primary care pediatric practice.

The primary aim is to compare the effectiveness of these two treatments in reducing body mass index (BMI) at 12 months. Secondary aims will compare impact of the treatments on reduction of risk factors related to cardiovascular disease and diabetes, including lipids, glucose and insulin, waist circumference, blood pressure, and measures of appetite. Further, the effectiveness of these two treatments in reducing BMI at 15 and 18 months will also be analyzed. Training aims will be met through collaboration with Lincoln University to set up undergraduate summer internships, graduate assistantships, and faculty development. Other methods for achieving the objectives of the Center include: a) establishing a multidisciplinary advisory board consisting of parents, providers, and researchers; b) providing clinical training in obesity treatment for doctors, nurses, dieticians, and behavioral interventionists at our collaborating institutions (CHOP and GHS); c) making all protocols and materials culturally sensitive to the populations they serve; and d) carrying out treatment development activities to tailor the manuals for Latino youth and their families.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adolescents
* Age 12 to 16 years
* Body Mass Index (BMI) of 28 kg/m2
* Adolescent expresses desire to lose weight
* Parent willing to participate
* Live within 40 minutes from study clinic at CHOP or 60 minutes at Geisinger

Exclusion Criteria:

* Uncontrolled hypertension (blood pressure > 140/90 mm HG)
* Diabetes mellitus (fasting glucose > 126 mg/dl)
* Any serious uncontrolled medical disorder that would complicate participation in a weight loss program
* Bipolar disorder or psychosis (depression ok if adolescent is receiving treatment)
* Use of any medication affecting body weight, appetite or metabolism within 30 days prior to the start of treatment
* Positive pregnancy test at medical evaluation

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 173 (Actual)
Dates: Start 2006-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Percentage change in initial body mass index (BMI) at 12 months | 12 months

SECONDARY OUTCOMES:
Compare mean reduction in percentage of initial BMI in the two treatments within each ethnic group/site (CHOP: urban African American adolescents and GHS: rural Caucasian adolescents | 12 months
Compare the effectiveness of the two treatment approaches on improving risk factors for cardiovascular disease and diabetes (Total, HDL, and LDL cholesterol, triglycerides, glucose, insulin, and blood pressure) and on improving liver function | 12 months
Compare mean reduction in percentage of initial BMI in each treatment group at month 6 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert I Berkowitz, MD, Principal Investigator — Children's Hospital of Philadelphia and University of Pennsylvania